CLINICAL TRIAL: NCT05226507
Title: A Phase 1 Clinical Study of NXP800 in Subjects With Advanced Cancers and Expansion in Subjects With Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nuvectis Pharma, Inc. (Industry)
Collaborators: Gynecologic Oncology Group Foundation (Unknown); The European Network for Gynaecological Oncological Trial groups (ENGOT) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NXP800-101; ENGOT-GYN5/GTG-UK/NXP800-101 (Other: ENGOT); GOG-3087 (Other: GOG Foundation)
Record Dates: First submitted 2022-01-13; First posted 2022-02-07 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor; Ovarian Cancer; Ovarian Clear Cell Carcinoma; Ovarian Clear Cell Tumor; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Endometrioid Tumor; ARID1A Gene Mutation
Keywords: Solid Tumor; Carcinoma; Neoplasms; Adenocarcinoma; ARID1a
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma; Neoplasms; Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: Part A dose escalation followed by Part B, expansion in ovarian cancers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part A: Dose Escalation (Experimental): Escalating doses of NXP800 administered orally once or twice daily.
  Interventions: Drug: NXP800
- Part B: Expansion in Ovarian Cancers Cohort 1 (Experimental): Subjects will be treated with NXP800 at 50 mg/day orally.
  Interventions: Drug: NXP800
- Part B: Expansion in Ovarian Cancers Cohort 2 (Experimental): Subjects will be treated with NXP800 at 75 mg/day orally.
  Interventions: Drug: NXP800

INTERVENTIONS:
Drug: NXP800 — NXP800 is an anti-neoplastic, oral small molecule.

SUMMARY:
The purpose of the dose escalation phase is to evaluate the safety profile of escalating doses and dose schedules of NXP800. In the expansion phase the preliminary efficacy in subjects with ARID1a mutated ovarian clear cell and ovarian endometrioid cancers will be estimated.

DETAILED DESCRIPTION:
Part A of the study is a dose escalation by cohort study of NXP800 administered to patients with advanced cancers. The study will identify the maximum tolerated dose (MTD) and propose dose and dose schedules for future studies.

In Part B doses selected in Part A are administered to patients with platinum-resistant, ARID1a-mutated ovarian carcinoma.

ELIGIBILITY:
Part A Inclusion Criteria:

* Provide written informed consent.
* 18 years old or older.
* Life expectancy of at least 12 weeks.
* Histologically- or cytologically-confirmed, advanced, metastatic, and/or progressive solid tumors for whom there is no authorized or effective therapy available, or for whom such therapies are considered inappropriate by the Investigator (in Part B, subjects with specific cancer types will be enrolled; Specific criteria will be introduced in a protocol amendment).
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.

Part A Exclusion Criteria:

* Radiotherapy (except for palliative reasons), endocrine therapy, chemotherapy, or investigational agent within 28 days, (42 days for nitrosoureas, mitomycin-C) of first dose of NXP800. Subjects can continue to receive bisphosphonates due to metastatic bone disease or GnRH agonists if they have prostate cancer.
* Ongoing toxic manifestations of previous treatments > Grade 2.
* Subjects with treated brain metastases are eligible if there is no evidence of progression for at least 28 days after central nervous system (CNS) directed treatment, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT] scan) during the Screening period.
* Female subjects who can become pregnant (or are already pregnant or lactating).
* Male subjects with partners of childbearing potential (unless they agree to take measures not to father children by using a barrier method of contraception (condom plus spermicide) or to sexual abstinence).

Part B Inclusion Criteria:

* Provide written informed consent.
* 18 years old or older.
* Subjects with the following ARID1a mutated, ovarian/fallopian tube/primary peritoneal cancer histologies (ARID1a mutation status determined by a DNA-based Next Generation Sequencing test):

  * Clear cell ovarian carcinoma (≥ 50% clear cell carcinoma with no serous differentiation)
  * Endometrioid ovarian carcinoma
* Subjects must have disease progression within 6 months (182 days) from completion of platinum-based therapy (6 months should be calculated from the date of the last administered dose of platinum therapy to the date of radiographic imaging showing progression)
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
* Subjects with a BRCA mutation must have received prior treatment with a PARP inhibitor.
* Subjects must have received at least 1 but not more than 3 prior systemic lines of anticancer therapy, including at least 1 line of therapy containing bevacizumab.

  * Adjuvant + neoadjuvant are considered one line of therapy
  * Maintenance therapy (i.e., bevacizumab, PARP inhibitors) will be considered as part of the preceeding line of therapy and are not counted independently.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Subjects must have a sufficient archival Formalin-Fixed Paraffin-Embedded (FFPE) tissue specimen, or be willing to consent to a fresh tissue biopsy during the study.

Part B Exclusion Criteria:

* Subjects with disease that did not respond to, or has progressed during or within 4 weeks of the last dose of first-line platinum containing chemotherapy.
* Radiotherapy (except for palliative reasons), endocrine therapy, chemotherapy, or investigational agent within 28 days, (42 days for nitrosoureas, mitomycin-C) of first dose of NXP800.
* Ongoing toxic manifestations of previous treatments > Grade 2, with the exception of alopecia.
* Subjects with treated brain metastases are eligible if there is no evidence of progression for at least 12 weeks while off corticosteroids after central nervous system (CNS) directed treatment, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT] scan) during the Screening period.
* Female subjects who can become pregnant (or are already pregnant or lactating).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Part B is enrolling ovarian cancer patients.
Enrollment: 45 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Part A: Number of patients with treatment related adverse events, clinical laboratory abnormalities, dose limiting toxicities | Day 28
Part B: Estimates of disease response by RECIST v 1.1 | Baseline to 30 days post last dose of NXP800
Part B: Number of patients with treatment related adverse events, and/or clinical laboratory abnormalities. | Baseline to 30 days post last dose of NXP800

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC) of NXP800 | First dose through Day 29
Maximum observed concentration (Cmax) of NXP800 | First dose through Day 29
Time to peak concentration (Tmax) of NXP800 | First dose through Day 29
Half-life (T1/2) of NXP800 | First dose through Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Udai Banerji, Prof, Principal Investigator — Institute of Cancer Research, Royal Marsden Foundation Trust; Susana Banerjee, Dr, Principal Investigator — Institute of Cancer Research, Royal Marsden NHS Foundation Trust
Locations (22):
- United States (19):
  - Honor Health, Phoenix, Arizona
  - UC San Diego Health - Moores Cancer Center, La Jolla, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale Gynecologic Oncology, New Haven, Connecticut
  - Florida Cancer Specialists South, Fort Myers, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Florida Cancer Specialists Research North, St. Petersburg, Florida
  - Florida Cancer Specialists Research East, West Palm Beach, Florida
  - University of Iowa, Iowa City, Iowa
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Women's Cancer Care Associates, Albany, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - Oncology Associates of Oregon, Eugene, Oregon
  - Sidney Kimmel Cancer Center, Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Texas Oncology, Fort Worth, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
- United Kingdom (3):
  - Royal Marsden Hospital, Sutton, Sutton Surrey
  - Addenbrookes Hospital, Cambridge
  - The Beatson West of Scotland Cancer Centre, Glasgow